CLINICAL TRIAL: NCT07181356
Title: Effects of Long-term Remote Ischemic Preconditioning on Clinical Outcome in Patients With Acute Myocardial Infarction
Acronym: L-RICP-AMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenanICE202105
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with acute myocardial infarction on admission were immediately assigned to the experimental group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group1（RIPerC+RIPC） (Experimental): Remote ischemic PERconditioning was initiated immediately after the diagnosis of acute myocardial infarction， and Remote ischemic PREconditioning was performed daily after discharge
  Interventions: Other: RIPerC; Other: RIPC
- Experimental Group2（RIPerC） (Experimental): Remote ischemic PERconditioning was initiated immediately after the diagnosis of acute myocardial infarction
  Interventions: Other: RIPerC
- Control group (No Intervention): A group of patients who received conventional treatment without any additional intervention

INTERVENTIONS:
Other: RIPerC — Each 40 minutes treatment time, 10 minutes as a cycle (cuff inflated to 200 mmHg and maintained for 5 minutes, then deflated for 5 minutes to start the next cycle), a total of 4 cycles
  Arms: Experimental Group1（RIPerC+RIPC）; Experimental Group2（RIPerC）
Other: RIPC — Each 40 minutes treatment time, 10 minutes as a cycle (cuff inflated to 200 mmHg and maintained for 5 minutes, then deflated for 5 minutes to start the next cycle), a total of 4 cycles
  Arms: Experimental Group1（RIPerC+RIPC）

SUMMARY:
At present, there are 290 million cardiovascular patients in China, including 11 million patients with coronary heart disease. Remote ischemic preconditioning(RIPC) may play an effective endogenous cardiac protection.This study will explore whether long-term use of RIPC in patients with AMI after PCI and non interventional therapy can reduce the incidence of major adverse cardiovascular cerebrovascular events(MACCE) and improve clinical outcomes and long-term prognosis.

DETAILED DESCRIPTION:
A total of 2146 patients with AMI are expected included as the research objects and randomly divided into experimental group and control group with 1073 cases in each group. After admission, Patients in the experimental group received everyday RIPC of upper limbs to the end of follow-up.The control group is a blank control and undergoes conventional medical procedures. Routine blood indexes, ultrasound, electrocardiogram, were detected On the day of admission. 12 months post- discharge, the incidence of MACCE(include Cardiovascular death, non-fatal acute myocardial infarction, stent thrombosis, revascularization, stroke, admission due to heart failure and the above composite events were independent components) and Poce(All deaths, all strokes, all myocardial infarction, or all revascularization events)will recorded by telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction were diagnosed in accordance with the criteria of the "Global Unified Definition of Fourth Myocardial Infarction"

Exclusion Criteria:

* The patients could not tolerate RIPC or RIPerC
* Aortic dissection, coronary artery aneurysm, coronary artery fistula and other systemic organic diseases
* The uncontrolled systolic blood pressure and diastolic blood pressure of severe hypertension were 180 mmHg and 120 mmHg respectively
* severe liver dysfunction (bilirubin > 20 mmol / L, prothrombin time > 2.0 ratio)
* Severe renal insufficiency (GFR < 30 ml / min / 1.73 m2);
* patients taking nicorandil and other drugs affecting microcirculation
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2146 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of MACCEs | 12 months after discharge
  MACCE(include Cardiovascular death, non-fatal acute myocardial infarction, revascularization, stroke, admission due to heart failure )

SECONDARY OUTCOMES:
Rate of Cardiovascular death events | 12 months after discharge
  Rate of Cardiovascular death events
Rate of non-fatal acute myocardial infarction events | 12 months after discharge
  Rate of non-fatal acute myocardial infarction events
Rate of revascularization events | 12 months after discharge
  Rate of revascularization events
Rate of stroke events | 12 months after discharge
  Rate of stroke events
Rate of admission due to heart failure events | 12 months after discharge
  Rate of admission due to heart failure events
Rate of all all-cause death events | 12 months after discharge
  Rate of all all-cause death events

CONTACTS AND LOCATIONS:
Overall Officials: Muwei LI, Ph.D, Study Chair — Fuwai Central China of Cardiovascular Hospital
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China